CLINICAL TRIAL: NCT02669706
Title: Assessment of the Safety and Intravenous Pentamidine for Pneumocystis Jirovecii Pneumonia in Patients With Hematologic Malignancies and Stem Cell Transplant Recipients.
Brief Title: Intravenous Pentamidine for Pneumocystis Jirovecii Pneumonia
Status: Completed | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Jennifer Anderson, PharmD, University of Illinois at Chicago
Other Study IDs: 2014-1000
Record Dates: First submitted 2016-01-25; First posted 2016-02-01 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Pentamidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IV pentamidine: Pentamidine 4mg/kg IV every month (maximum 300mg)
  Interventions: Drug: Pentamidine

INTERVENTIONS:
Drug: Pentamidine — Pentamidine is an antimicrobial medication given for prevention and treatment of Pneumocystis pneumonia (PJP) caused by Pneumocystis jirovecii
  Other Names: NebuPent; Pentam

SUMMARY:
The main objective of this study is to assess the safety of administering intravenous (IV) pentamidine for Pneumocystis jirovecii pneumonia (PJP) prophylaxis in adult inpatients with hematologic malignancies and stem cell transplant recipients. There will also be an assessment of patient satisfaction associated with intravenous pentamidine PJP prophylactic therapy.

DETAILED DESCRIPTION:
This study is a prospective, single arm study to assess safety of IV pentamidine for PJP prophylaxis. Patient satisfaction associated with IV pentamidine will also be assessed using a survey adapted from the validated Treatment Satisfaction Questionnaire for Medication (version 1.4).

Adult patients with a hematologic malignancy or who are receiving or have received a stem-cell transplant at the University of Illinois Hospitals and Clinics who have an indication for PJP prophylaxis therapy. They will receive intravenous pentamidine during their planned admissions for chemotherapy when they have an indication for and/or are due to receive pentamidine prophylaxis. These patients are outlined below in the inclusion criteria. Patients may or may not have received aerosolized or IV pentamidine prior to inclusion in the study.

Eligible patients will receive IV pentamidine during hospital admissions. Patients will be routinely monitored by nursing staff during and after the infusion. Nursing staff will monitor the systolic and diastolic blood pressure at baseline and one hour post infusion. Patients will also be monitored for nausea/vomiting. Patients who receive IV pentamidine will have anti-emetics available on call to use in the event that they become nauseous. Data will be collected on the type, grade, and incidence of adverse effects by research personnel.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Hematologic malignancy diagnosis or stem-cell transplant recipient
* Eligible for PJP prophylaxis therapy at time of enrollment as per institutional guidelines in compliance with NCCN guidelines. These patients include:
* Acute myeloid leukemia patients receiving induction and consolidation (first line and relapsed/refractory)
* Acute lymphoid leukemia patients receiving HyperCVAD/R (cyclophosphamide, vincristine, doxorubicin, dexamethasone, methotrexate, cytarabine, rituximab)
* Lymphoma patients receiving ICE (ifosfamide, carboplatin, etoposide), DA-R-EPOCH (dose-adjusted rituximab, etoposide, prednisone, vincristine, cyclophosphamide, doxorubicin), and other inpatient lymphoma regimens
* Patients receiving other inpatient chemotherapy regimens that are given on a monthly basis
* Patients who have received an allogeneic stem cell transplant
* Have given informed consent
* May have previously received inhaled or IV pentamidine

Exclusion Criteria:

* Pregnancy
* Prisoners
* Patients with a documented allergy or hypersensitivity to pentamidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of adult patients with hematologic malignancies and/or hematopoietic stem cell transplant recipients who have an indication for PJP prophylaxis with pentamidine. Further details are outlined in the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Safety of IV pentamidine for PJP prophylaxis | 1 year
  Safety will be assessed via analyzing the number of patients experiencing adverse effects, with their severity graded using CTCAE v4.0.

SECONDARY OUTCOMES:
Number of confirmed cases of PJP diagnosed | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Anderson, PharmD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Hospital and Health Sciences System, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Morris A, Norris KA. Colonization by Pneumocystis jirovecii and its role in disease. Clin Microbiol Rev. 2012 Apr;25(2):297-317. doi: 10.1128/CMR.00013-12. PMID 22491773
- [Background] Green H, Paul M, Vidal L, Leibovici L. Prophylaxis of Pneumocystis pneumonia in immunocompromised non-HIV-infected patients: systematic review and meta-analysis of randomized controlled trials. Mayo Clin Proc. 2007 Sep;82(9):1052-9. doi: 10.4065/82.9.1052. PMID 17803871
- [Background] Orgel E, Rushing T. Efficacy and tolerability of intravenous pentamidine isethionate for Pneumocystis jiroveci prophylaxis in a pediatric oncology population. Pediatr Infect Dis J. 2014 Mar;33(3):319-21. doi: 10.1097/INF.0000000000000044. PMID 24030353
- [Background] Sahoo RC. Adenosine deaminase in the diagnosis of tubercular pleural effusion--how far it is helpful. J Assoc Physicians India. 1992 Nov;40(11):772. No abstract available. PMID 1307553
- [Background] DeMasi JM, Cox JA, Leonard D, Koh AY, Aquino VM. Intravenous pentamidine is safe and effective as primary pneumocystis pneumonia prophylaxis in children and adolescents undergoing hematopoietic stem cell transplantation. Pediatr Infect Dis J. 2013 Sep;32(9):933-6. doi: 10.1097/INF.0b013e318292f560. PMID 23538522
- [Background] Kim SY, Dabb AA, Glenn DJ, Snyder KM, Chuk MK, Loeb DM. Intravenous pentamidine is effective as second line Pneumocystis pneumonia prophylaxis in pediatric oncology patients. Pediatr Blood Cancer. 2008 Apr;50(4):779-83. doi: 10.1002/pbc.21287. PMID 17635000
- [Derived] Sweiss K, Anderson J, Wirth S, Oh A, Quigley JG, Khan I, Saraf S, Mactal-Haaf C, Rondelli D, Patel P. A prospective study of intravenous pentamidine for PJP prophylaxis in adult patients undergoing intensive chemotherapy or hematopoietic stem cell transplant. Bone Marrow Transplant. 2018 Mar;53(3):300-306. doi: 10.1038/s41409-017-0024-1. Epub 2017 Dec 21. PMID 29269796